CLINICAL TRIAL: NCT00281450
Title: A Cluster Randomized Educational Intervention to Reduce Inappropriate Prescription Patterns for Elderly Patients in General Practice
Brief Title: An Intervention to Reduce Inappropriate Prescriptions for Elderly Patients in General Practice
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Jorund Straand, professor MD PhD, University of Oslo
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 850652
Record Dates: First submitted 2006-01-03; First posted 2006-01-24 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2005-12

CONDITIONS: Aged; Family Practice
MeSH Terms: interventions — Early Intervention, Educational

INTERVENTIONS:
Behavioral: Educational intervention — We developed a set of explicit criteria for pharmacological inappropriateness for Norwegian GPs' prescribing to elderly patients. The main purpose of the criteria was to serve as quality indicators during an educational intervention: the Prescription Peer Academic Detailing (Rx-PAD) Study, aimed at improving GPs' prescribing for elderly patients.

SUMMARY:
This study will explore the possible effect of a tailored educational intervention towards general practitioners, in order to reduce inappropriate prescription patterns for elderly patients > 70 years.

ELIGIBILITY:
Inclusion Criteria:

* General practitioner
* Specialist in general practice

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85836 (Actual)
Dates: Start 2006-01; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Changes in a set of predefined quality indicators measuring appropriateness of prescriptions for elderly out-patients | 1 year
  Prescription data for 1 year were retrospectively retrieved from the Norwegian Prescription Database (NorPD) and assessed in relation to 13 prescription quality indicators.

CONTACTS AND LOCATIONS:
Overall Officials: Sture Rognstad, MD, Principal Investigator — University of Oslo

REFERENCES:
- [Derived] Straand J, Fetveit A, Rognstad S, Gjelstad S, Brekke M, Dalen I. A cluster-randomized educational intervention to reduce inappropriate prescription patterns for elderly patients in general practice--The Prescription Peer Academic Detailing (Rx-PAD) study [NCT00281450]. BMC Health Serv Res. 2006 Jun 11;6:72. doi: 10.1186/1472-6963-6-72. PMID 16764734